CLINICAL TRIAL: NCT01680016
Title: A Phase IIIb, Randomized, Open-label Study Comparing Two Different Rabies Vaccine Post-exposure Schedules (Zagreb 2-1-1 and Rabipur® Essen 1-1-1-1-1) in Chinese Children and Older Adults
Brief Title: A Randomized, Open-label Study Comparing Two Different Rabies Vaccine Schedules in Chinese Children and Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V49_24
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-04

CONDITIONS: Rabies
Keywords: Rabies virus, postexposure, vaccine schedule, children, older adults
MeSH Terms: conditions — Rabies | interventions — hemoglobin A2 Zagreb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Zagreb(≥6 to ≤17 Years) (Experimental)
  Interventions: Biological: Zagreb
- Zagreb(≥51 Years) (Experimental)
  Interventions: Biological: Zagreb
- Essen(≥6 to ≤17 Years) (Active Comparator)
  Interventions: Biological: Essen
- Essen(≥51 Years) (Active Comparator)
  Interventions: Biological: Essen

INTERVENTIONS:
Biological: Zagreb — Subjects received Zagreb schedule (2-1-1) i.e. 4 vaccinations of Rabipur at days 1 , 8 and 22
  Arms: Zagreb(≥51 Years); Zagreb(≥6 to ≤17 Years)
Biological: Essen — Subjects received Essen schedule (1-1-1-1-1) i.e. 5 vaccinations of Rabipur at days 1, 4, 8, 15 and 29
  Arms: Essen(≥51 Years); Essen(≥6 to ≤17 Years)

SUMMARY:
This study was designed to evaluate the safety and immunogenicity of two simulated postexposure rabies vaccination schedules (Zagreb 2-1-1 and Essen 1-1-1-1-1) in Chinese children and older adults.

DETAILED DESCRIPTION:
This study was designed to evaluate the safety and immunogenicity of Rabipur Zagreb (2-1-1) and Rabipur Essen (1-1-1-1-1) simulated post exposure vaccination schedules in Chinese children and older adults. Subjects randomized to Group 1 (Zagreb) will receive 4 doses of rabies vaccine Day 1 (2 doses), and on Day 8 and Day 22. Subjects randomized to Group 2 (Essen) will receive 5 doses of rabies vaccine on Days 1, 4, 8, 15, and 29. First vaccine will be administered on study Day 1.

240 children and 400 older adults, a total of 640, is planned to be enrolled into the study. Subjects will be divided further into age subsets of equal numbers within each age cohort (children: 6 to 11 years of age and 12 to 17 years of age; older adults: 51 to 60 years of age and 61 years of age and older. Within each age subset, subjects will be assigned randomly in a 1:1 ratio.

The primary objective is to establish the non-inferiority of the Rabipur Zagreb (2-1-1) schedule relative to the conventional Rabipur Essen (1-1-1-1-1) schedule based on geometric mean titers (GMC), and the secondary objective is to assess the percent of subjects with rabies virus neutralizing titer ≥ 0.5 IU/mL 14 days after the first vaccinations (study Day 15) for each schedule and age cohort

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 6-17 years of age and 51 years of age or older
* Individuals who were in good health
* Provided consent, complied with study procedures and duration of follow-up

Exclusion Criteria:

* Contraindications to vaccination with rabies vaccine
* Body temperature ≥37.5◦C (axillary) within 3 days of intended study vaccination
* Known hypersensitivity to the components of the vaccine
* Previously received any rabies vaccine or immune globulin
* Previous or planned treatment with antimalarial medications
* History of psychiatric disease, immune disorder, bleeding disorder, drug/alcohol abuse within the past 2 years, malignancy
* Female subjects who were pregnant or unwilling to practice acceptable birth control methods
* Individuals enrolled or plans to enroll in another investigational trial

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Mengshan Center for Disease Prevention and Control (CDC), Mengshan, Guangxi, China

REFERENCES:
- [Derived] Li R, Li Y, Wen S, Wen H, Nong Y, Mo Z, Xie F, Pellegrini M. Immunogenicity and safety of purified chick-embryo cell rabies vaccine under Zagreb 2-1-1 or 5-dose Essen regimen in Chinese children 6 to 17 years old and adults over 50 years: a randomized open-label study. Hum Vaccin Immunother. 2015;11(2):435-42. doi: 10.4161/21645515.2014.994460. PMID 25692350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Mengshan CDC
Pre-assignment Details: All enrolled subjects were included in the trial
Groups:
- Zagreb(≥6 to ≤17 Years): ≥6 to ≤17 years-old subjects received Zagreb schedule (2-1-1) i.e. 4 vaccinations of Rabipur at days 1, 8 and 22
- Essen(≥6 to ≤17 Years): ≥6 to ≤17 years-old subjects received Essen schedule (1-1-1-1-1) i.e. 5 vaccinations of Rabipur at days 1, 4, 8, 15 and 29
- Zagreb(≥51 Years): ≥51 years-old subjects received Zagreb schedule (2-1-1) i.e. 4 vaccinations of Rabipur at days 1 , 8 and 22
- Essen(≥51 Years): ≥51 years-old subjects received Essen schedule (1-1-1-1-1) i.e. 5 vaccinations of Rabipur at days 1, 4, 8, 15 and 29
Period: Overall Study
Arm/Group | Zagreb(≥6 to ≤17 Years) | Essen(≥6 to ≤17 Years) | Zagreb(≥51 Years) | Essen(≥51 Years)
Started | 121 | 122 | 201 | 200
Completed | 115 | 114 | 196 | 195
Not Completed | 6 | 8 | 5 | 5
Not completed — Adverse Event | 0 | 0 | 1 | 4
Not completed — The Subject went out of The Trial | 1 | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 7 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled set:All subjects who had signed an informed consent, undergone screening procedure(s) and were randomized
Groups:
- Zagreb: Zagreb schedule (2-1-1) i.e. 4 vaccinations of Rabipur at days 1 , 8 and 22
- Essen: Essen schedule (1-1-1-1-1) i.e. 5 vaccinations of Rabipur at days 1, 4, 8, 15 and 29
- Total: Total of all reporting groups
Arm/Group | Zagreb | Essen | Total
Number analyzed (Participants) | 322 | 322 | 644
Age, Continuous [Mean (Standard Deviation); unit: years]
  Children (≥6 to ≤17 Years) | 11 (3.0) | 10.8 (2.9) | 10.9 (3.0)
  Older Adults (≥51 Years) | 62.1 (6.5) | 61.9 (6.8) | 62.0 (6.6)
Sex/Gender, Customized [Number; unit: Subjects]
  Female (≥6 to ≤17 Years) | 49 | 76 | 125
  Male (≥6 to ≤17 Years) | 72 | 46 | 118
  Female (≥51 Years) | 118 | 123 | 241
  Male (≥51 Years) | 83 | 77 | 160

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority in Immune Response of the Zagreb Postexposure Schedule of Rabipur to That of the Conventional Essen Postexposure Schedule of Rabipur as Measured by GMC of RVNA Titer 14 Days After First Vaccination in Children Aged ≥6 to ≤17 Years.
Description: Immunogenicity was measured as the geometric mean concentrations (GMCs) of rabies virus neutralizing antibody (RVNA) titer , evaluated using the rapid fluorescent focus inhibition test, before vaccination and 14 days after first vaccination of Rabipur as per Zagreb (2-1-1) and Essen (1-1-1-1-1) postexposure schedule.
Time Frame: Before vaccination (day 1) and 14 days after first vaccination (day 15)
Population: Analysis was done on the per-protocol (PP) set, i.e. the subjects who received the vaccine correctly; provided evaluable serum samples at the relevant time points; and had no major protocol violations as defined prior to analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Zagreb(≥6 to ≤17 Years) | Essen(≥6 to ≤17 Years)
Number analyzed (Participants) | 114 | 110
IU/mL
  Day 1 | 0.052 [0.048 to 0.056] | 0.054 [0.05 to 0.058]
  Day 15 | 12 [10 to 14] | 14 [12 to 16]
Statistical Analysis 1: Comparison: Zagreb(≥6 to ≤17 Years) vs Essen(≥6 to ≤17 Years); To demonstrate noninferiority in immune response of the Zagreb post-exposure schedule of Rabipur to that of the conventional Essen post-exposure schedule at day 15 in children aged ≥6 to ≤17 years; Test type: Non-Inferiority or Equivalence — Noninferiority was achieved if the lower limit of the two-sided 95% CI around the observed ratio of GMCs between the groups (GMCGroup Zagreb / GMCGroup Essen) was greater than 0.5; ANOVA; Ratio of GMCs between two groups(Day 15) = 0.84, 95% CI 2-sided [0.69 to 1.02]

2. Primary Outcome: Non-inferiority in Immune Response of the Zagreb Postexposure Schedule of Rabipur to That of the Conventional Essen Postexposure Schedule of Rabipur as Measured by GMC of RVNA Titer 14 Days After the First Vaccination in Older Adults Aged ≥51 Years
Description: Immunogenicity was measured as the GMCs of Rabies Virus Neutralizing Antibody (RVNA) titer , evaluated using the rapid fluorescent focus inhibition test, before vaccination and 14 days after first vaccination of Rabipur as per Zagreb (2-1-1) and Essen (1-1-1-1-1) postexposure schedule.
Time Frame: Before vaccination (day 1) and 14 days after first vaccination (day 15).
Population: Analysis was done on the PP set.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Zagreb(≥51 Years) | Essen(≥51 Years)
Number analyzed (Participants) | 190 | 188
IU/mL
  Day 1 | 0.057 [0.052 to 0.063] | 0.06 [0.055 to 0.066]
  Day 15 | 8.57 [7.34 to 10] | 7.89 [6.75 to 9.21]
Statistical Analysis 1: Comparison: Zagreb(≥51 Years) vs Essen(≥51 Years); To demonstrate noninferiority in immune response of the Zagreb post-exposure schedule of Rabipur to that of the conventional Essen post-exposure schedule at day 15 in older adults aged ≥51 years; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of GMCs between two groups(Day 15) = 1.09, 95% CI 2-sided [0.87 to 1.35]

3. Secondary Outcome: Percentages of Children With RVNA Titers ≥0.5 IU/mL 14 Days After First Vaccination of Rabipur
Description: Immunogenicity was measured as the percentages of subjects who achieved RVNA titers ≥0.5 IU/mL, 14 days after first vaccination of Rabipur as per Zagreb (2-1-1) and Essen (1-1-1-1-1) postexposure schedule.
Time Frame: Before vaccination (day 1) and 14 days after first vaccination (day 15).
Population: For the analysis of this outcome measure children aged ≥6 to ≤17 years were divided into two subgroups, i.e. ≥6 to ≤11 years and ≥12 to ≤17 years. Analysis was done on the PP set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- Zagreb(≥6 to ≤11 Years): ≥6 to ≤11 years-old subjects received Zagreb schedule (2-1-1) i.e. 4 vaccinations of Rabipur at days 1 , 8 and 22
- Essen(≥6 to ≤11 Years): ≥6 to ≤11 years-old subjects received Essen schedule (1-1-1-1-1) i.e. 5 vaccinations of Rabipur at days 1, 4, 8, 15 and 29
- Zagreb(≥12 to ≤17 Years): ≥12 to ≤17 years-old subjects received Zagreb schedule (2-1-1) i.e. 4 vaccinations of Rabipur at days 1 , 8 and 22
- Essen(≥12 to ≤17 Years): ≥12 to ≤17 years-old subjects received Essen schedule (1-1-1-1-1) i.e. 5 vaccinations of Rabipur at days 1, 4, 8, 15 and 29
- Zagreb( ≥6 to ≤17 Years): ≥6 to ≤17 years-old subjects received Zagreb schedule (2-1-1) i.e. 4 vaccinations of Rabipur at days 1 , 8 and 22
Arm/Group | Zagreb(≥6 to ≤11 Years) | Essen(≥6 to ≤11 Years) | Zagreb(≥12 to ≤17 Years) | Essen(≥12 to ≤17 Years) | Zagreb( ≥6 to ≤17 Years) | Essen(≥6 to ≤17 Years)
Number analyzed (Participants) | 58 | 56 | 56 | 54 | 114 | 110
Percentages of subjects
  Day 1(58,56,56,54,114,110) | 0 [0 to 6] | 2 [0.045 to 10] | 0 [0 to 6] | 4 [0 to 13] | 0 [0 to 3] | 3 [1 to 8]
  Day 15(58,56,56,54,114, 110) | 100 [94 to 100] | 100 [94 to 100] | 100 [94 to 100] | 100 [93 to 100] | 100 [97 to 100] | 100 [97 to 100]

4. Secondary Outcome: Percentages of Older Adults With RVNA Titers ≥0.5 IU/mL 14 Days After First Vaccination of Rabipur
Description: as for outcome 3
Time Frame: Before vaccination (day 1) and 14 days after first vaccination (day 15).
Population: For the analysis of this outcome measure older adults aged ≥51 years were divided into two subgroups, i.e. ≥51 to ≤60 years and ≥61 years. Analysis was done on the PP set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- Zagreb(≥51 to ≤60 Years): ≥51 to ≤60 years-old subjects received Zagreb schedule (2-1-1) i.e. 4 doses of Rabipur at days 1 , 8 and 22
- Essen(≥51 to ≤60 Years): ≥51 to ≤60 years-old subjects received Essen schedule (1-1-1-1-1) i.e. 5 vaccinations of Rabipur at days 1, 4, 8, 15 and 29
- Zagreb(≥61 Years): ≥61 years-old subjects received Zagreb schedule (2-1-1) i.e. 4 doses of Rabipur at days 1 , 8 and 22
- Essen(≥61 Years): ≥61 years-old subjects received Essen schedule (1-1-1-1-1) i.e. 5 vaccinations of Rabipur at days 1, 4, 8, 15 and 29
- Zagreb(≥51 Years): ≥51 years-old subjects received Zagreb schedule (2-1-1) i.e. 4 doses of Rabipur at days 1 , 8 and 22
Arm/Group | Zagreb(≥51 to ≤60 Years) | Essen(≥51 to ≤60 Years) | Zagreb(≥61 Years) | Essen(≥61 Years) | Zagreb(≥51 Years) | Essen(≥51 Years)
Number analyzed (Participants) | 93 | 93 | 97 | 95 | 190 | 188
Percentages of subjects
  Day 1(93,93,97,95,190,188) | 5 [2 to 12] | 4 [1 to 11] | 1 [0.026 to 6] | 4 [1 to 10] | 3 [1 to 7] | 4 [2 to 8]
  Day 15 (93,93,97,95,190, 188) | 100 [96 to 100] | 100 [96 to 100] | 99 [94 to 100] | 99 [94 to 100] | 99 [97 to 100] | 99 [97 to 100]

5. Secondary Outcome: Percentages of Children With RVNA Titers ≥0.5 IU/mL 42 Days After First Vaccination of Rabipur
Description: Immunogenicity was measured as the percentages of subjects who achieved RVNA titers ≥0.5 IU/mL, 42 days after first vaccination of Rabipur as per Zagreb (2-1-1) and Essen (1-1-1-1-1) postexposure schedule.
Time Frame: Before vaccination (day 1) and 42 days after first vaccination (day 43).
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Zagreb(≥6 to ≤11 Years) | Essen(≥6 to ≤11 Years) | Zagreb(≥12 to ≤17 Years) | Essen(≥12 to ≤17 Years) | Zagreb( ≥6 to ≤17 Years) | Essen(≥6 to ≤17 Years)
Number analyzed (Participants) | 57 | 56 | 56 | 55 | 113 | 111
Percentages of subjects
  Day 1(57,56,56,55,113,111) | 0 [0 to 6] | 2 [0.045 to 10] | 0 [0 to 6] | 4 [0 to 13] | 0 [0 to 3] | 3 [1 to 8]
  Day 43 (57,56,56,55,113,111) | 100 [94 to 100] | 100 [94 to 100] | 100 [94 to 100] | 100 [94 to 100] | 100 [97 to 100] | 100 [97 to 100]

6. Secondary Outcome: Percentages of Older Adults With RVNA Titers ≥0.5 IU/mL 42 Days After First Vaccination of Rabipur
Description: as for outcome 5
Time Frame: Before vaccination (day 1) and 42 days after first vaccination (day 43).
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Zagreb(≥51 to ≤60 Years) | Essen(≥51 to ≤60 Years) | Zagreb(≥61 Years) | Essen(≥61 Years) | Zagreb(≥51 Years) | Essen(≥51 Years)
Number analyzed (Participants) | 92 | 90 | 96 | 93 | 188 | 183
Percentages of subjects
  Day 1(92,90,96,93,188,183) | 5 [2 to 12] | 4 [1 to 11] | 1 [0.026 to 6] | 4 [1 to 11] | 3 [1 to 7] | 4 [2 to 8]
  Day 43 (92,90,96,93,188,183) | 100 [96 to 100] | 100 [96 to 100] | 100 [96 to 100] | 100 [96 to 100] | 100 [98 to 100] | 100 [98 to 100]

7. Primary Outcome: Number of Children Who Reported Solicited Local and Systemic Adverse Events After Any Vaccination of Rabipur
Description: Safety was assessed as the number of children who reported solicited local and systemic adverse events from day 1 up to and including day 7 after any vaccination of Rabipur as per Zagreb (2-1-1) and Essen (1-1-1-1-1) postexposure schedule.
Time Frame: Days 1 to 7 postvaccination
Population: Analysis was done on the safety set, i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: Subjects
Arm/Group | Zagreb(≥6 to ≤11 Years) | Essen(≥6 to ≤11 Years) | Zagreb(≥12 to ≤17 Years) | Essen(≥12 to ≤17 Years) | Zagreb( ≥6 to ≤17 Years) | Essen(≥6 to ≤17 Years)
Number analyzed (Participants) | 60 | 59 | 61 | 60 | 121 | 119
Subjects
  Injection Site Erythema(N=59,58,60,60,119,118) | 2 | 1 | 0 | 0 | 2 | 1
  Injection Site Induration(N=59,58,60,60,119,118) | 1 | 0 | 1 | 0 | 2 | 0
  Injection Site Pain(N=59,58,60,60,119,118) | 21 | 18 | 24 | 29 | 45 | 47
  Nausea(N=59,58,60,60,119,118) | 2 | 4 | 5 | 6 | 7 | 10
  Myalgia(N=59,58,60,60,119,118) | 4 | 4 | 7 | 9 | 11 | 13
  Arthralgia(N=59,58,60,60,119,118) | 1 | 0 | 2 | 1 | 3 | 1
  Headache(N=59,58,60,60,119,118) | 4 | 4 | 7 | 6 | 11 | 10
  Fatigue(N=59,58,60,60,119,118) | 8 | 4 | 10 | 11 | 18 | 15
  Loss of Appetite(N=59,58,60,60,119,118) | 7 | 3 | 7 | 7 | 14 | 10
  Body Temp. (≥38°C)(N=59,58,60,60,119,118) | 6 | 3 | 2 | 0 | 8 | 3
  Low Grade Fever(N=59,58,60,60,119,118) | 6 | 7 | 11 | 11 | 17 | 18
  Medium Grade Fever(N=59,58,60,60,119,118) | 9 | 5 | 4 | 2 | 13 | 7
  High Grade Fever(N=59,58,60,60,119,118) | 0 | 0 | 0 | 0 | 0 | 0
  Analge,Antipyr Used(N=59,58,60,60,119,118) | 7 | 4 | 4 | 4 | 11 | 8

8. Primary Outcome: Number of Older Adults Who Reported Solicited Local and Systemic Adverse Events After Any Vaccination of Rabipur
Description: Safety was assessed as the number of subjects who reported solicited local and systemic adverse events from day 1 up to and including day 7 after any vaccination of Rabipur as per Zagreb (2-1-1) and Essen (1-1-1-1-1) postexposure schedule.
Time Frame: Days 1 to 7 postvaccination
Population: Analysis was done on the safety set
Measure: Number; unit: Subjects
Arm/Group | Zagreb(≥51 to ≤60 Years) | Essen(≥51 to ≤60 Years) | Zagreb(≥61 Years) | Essen(≥61 Years) | Zagreb(≥51 Years) | Essen(≥51 Years)
Number analyzed (Participants) | 100 | 100 | 100 | 100 | 200 | 200
Subjects
  Injection Site Erythema(N=98,100,99,100,197,200) | 1 | 1 | 0 | 2 | 1 | 3
  Injection Site Induration(N=98,100,99,100,197,200) | 1 | 1 | 0 | 0 | 1 | 1
  Injection Site Pain(N=98,100,99,100,197,200) | 9 | 12 | 9 | 10 | 18 | 22
  Nausea(N=98,100,99,100,197,200) | 1 | 0 | 1 | 2 | 2 | 2
  Myalgia(N=98,100,99,100,197,200) | 0 | 0 | 0 | 2 | 0 | 2
  Arthralgia(N=98,100,99,100,197,200) | 0 | 2 | 3 | 1 | 3 | 3
  Headache(N=98,100,99,100,197,200) | 4 | 2 | 3 | 6 | 7 | 8
  Fatigue(N=98,100,99,100,197,200) | 3 | 4 | 6 | 3 | 9 | 7
  Loss of Appetite(N=98,100,99,100,197,200) | 0 | 1 | 0 | 1 | 0 | 2
  Body Temp.(≥38°C)(N=98,100,99,100,197,200) | 0 | 1 | 5 | 4 | 5 | 5
  Low Grade Fever(N=98,100,99,100,197,200) | 3 | 5 | 3 | 6 | 6 | 11
  Medium Grade Fever(N=98,100,99,100,197,200) | 1 | 2 | 5 | 6 | 6 | 8
  High Grade Fever(N=98,100,99,100,197,200) | 0 | 0 | 1 | 0 | 1 | 0
  Analgesic,Antipyretic use(N=98,100,99,100,197,200) | 6 | 6 | 7 | 9 | 13 | 15

9. Secondary Outcome: GMCs of RVNA Titer 42 Days After First Vaccination in Children.
Description: Immunogenicity was measured as the GMCs of RVNA titers, evaluated using the rapid fluorescent focus inhibition test, before vaccination and 42 days after first vaccination of Rabipur as per Zagreb (2-1-1) and Essen (1-1-1-1-1) postexposure schedule.
Time Frame: Before vaccination (day 1) and 42 days after first vaccination (day 43)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Concentration (IU/mL)
Arm/Group | Zagreb(≥6 to ≤11 Years) | Essen(≥6 to ≤11 Years) | Zagreb(≥12 to ≤17 Years) | Essen(≥12 to ≤17 Years) | Zagreb( ≥6 to ≤17 Years) | Essen(≥6 to ≤17 Years)
Number analyzed (Participants) | 57 | 56 | 56 | 55 | 113 | 111
Concentration (IU/mL)
  Day 1(N=57,56,56,55,113,111) | 0.054 [0.048 to 0.06] | 0.053 [0.048 to 0.059] | 0.05 [0.046 to 0.055] | 0.055 [0.05 to 0.06] | 0.052 [0.048 to 0.056] | 0.054 [0.05 to 0.058]
  Day 43(N=57,56,56,55,113,111) | 13 [11 to 15] | 24 [20 to 29] | 13 [11 to 16] | 23 [19 to 28] | 13 [11 to 15] | 24 [21 to 27]

10. Secondary Outcome: GMCs of RVNA Titer 42 Days After the First Vaccination in Older Adults.
Description: as for outcome 9
Time Frame: Before vaccination (day 1) and 42 days after first vaccination (day 43)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Concentration (IU/ml)
Arm/Group | Zagreb(≥51 to ≤60 Years) | Essen(≥51 to ≤60 Years) | Zagreb(≥61 Years) | Essen(≥61 Years) | Zagreb(≥51 Years) | Essen(≥51 Years)
Number analyzed (Participants) | 92 | 90 | 96 | 93 | 188 | 183
Concentration (IU/ml)
  Day 1(92,90,96,93,188,183) | 0.063 [0.054 to 0.074] | 0.06 [0.052 to 0.07] | 0.052 [0.047 to 0.058] | 0.06 [0.054 to 0.068] | 0.057 [0.052 to 0.063] | 0.06 [0.055 to 0.066]
  Day 43(92,90,96,93,188,183) | 12 [9.36 to 15] | 16 [13 to 20] | 12 [9.39 to 15] | 11 [8.67 to 14] | 12 [10 to 14] | 13 [11 to 16]

11. Primary Outcome: Number of Children Who Reported Unsolicited Adverse Events (AEs)
Description: The safety of Rabipur was assessed in terms of subjects(Children) exposed to study vaccine who reported all Unsolicited AEs (including serious adverse events [SAE]s and AEs leading to subject withdrawal) from V1/day 1 (postvaccination) through V7/study termination day 43.
Time Frame: From V1/day 1 (postvaccination) through V7/study termination day 43
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Zagreb(≥6 to ≤17 Years) | Essen(≥6 to ≤17 Years)
Number analyzed (Participants) | 121 | 119
Subjects
  Any unsolicited AEs | 26 | 28
  At least possibly related unsolicited AEs | 9 | 6
  Serious AEs | 0 | 0
  At least possibly related Serious AEs | 0 | 0
  Death | 0 | 0
  Premature withdrawals due to AEs | 0 | 0

12. Primary Outcome: Number of Older Adults Who Reported Unsolicited Adverse Events (AEs)
Description: The safety of Rabipur was assessed in terms of subjects(Older Adults) exposed to study vaccine who reported all Unsolicited AEs (including serious adverse events [SAE]s and AEs leading to subject withdrawal) from V1/day 1 (postvaccination) through V7/study termination day 43.
Time Frame: from V1/day 1 (postvaccination) through V7/study termination day 43
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Zagreb(≥51 Years) | Essen(≥51 Years)
Number analyzed (Participants) | 200 | 200
Subjects
  Any unsolicited AEs | 36 | 39
  At least possibly related unsolicited AEs | 5 | 15
  Serious AEs | 1 | 0
  At least possibly related Serious AEs | 0 | 0
  Death | 0 | 0
  Premature withdrawals due to AEs | 1 | 4

ADVERSE EVENTS:
Time Frame: Whole study period (From day 1 to day 43)
Description: Serious adverse events (SAEs) were collected from day 1 to study termination (day 43).The safety analysis was performed in all exposed set -All subjects in the Enrolled Set who received a study vaccination
Groups:
- Zagreb(≥6 to ≤17 Years): ≥6 to ≤17 years-old subjects received Zagreb schedule (2-1-1) i.e. 4 doses of Rabipur at days 1 , 8 and 22
- Essen(≥6 to ≤17 Years): ≥6 to ≤17 years-old subjects received Essen schedule (1-1-1-1-1) i.e. 5 doses of Rabipur at days 1, 4, 8, 15 and 29
- Essen(≥51 Years): ≥51 years-old subjects received Essen schedule (1-1-1-1-1) i.e. 5 doses of Rabipur at days 1, 4, 8, 15 and 29
Arm/Group | Zagreb(≥6 to ≤17 Years) | Essen(≥6 to ≤17 Years) | Zagreb(≥51 Years) | Essen(≥51 Years)
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/119 | 1/200 | 0/200
Other Adverse Events (participants affected / at risk) | 64/121 | 63/119 | 19/200 | 24/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zagreb(≥6 to ≤17 Years) (N=121) | Essen(≥6 to ≤17 Years) (N=119) | Zagreb(≥51 Years) (N=200) | Essen(≥51 Years) (N=200)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zagreb(≥6 to ≤17 Years) (N=121) | Essen(≥6 to ≤17 Years) (N=119) | Zagreb(≥51 Years) (N=200) | Essen(≥51 Years) (N=200)
Fatigue (General disorders) | 18 | 15 | 9 | 7
Injection Site Pain (General disorders) | 48 | 50 | 19 | 24
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 13 | 5 | 6
Headache (Nervous system disorders) | 11 | 10 | 8 | 9
Nausea (Gastrointestinal disorders) | 7 | 10 | 4 | 2
Injection Site Erythema (General disorders) | 8 | 2 | 1 | 5
Pyrexia (General disorders) | 8 | 3 | 5 | 7
Decreased Appetite (Metabolism and nutrition disorders) | 14 | 10 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 13 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial